CLINICAL TRIAL: NCT07307495
Title: Effect of Postoperative Analgesia of Oliceridine Fumarate for Gastrointestinal Function Recovery in Patients Undergoing Lumbar Spine Surgery:A Prospective, Multicenter, Double-blind,Randomized Controlled Study
Brief Title: Effect of Postoperative Analgesia of Oliceridine Fumarate for Gastrointestinal Function Recovery in Patients Undergoing Lumbar Spine Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20252506-F-2
Record Dates: First submitted 2025-11-18; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Oliceridine Fumarate
Keywords: lumbar spine surgery; gastrointestinal function recovery
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine Group (Experimental): Oliceridine Patient-Controlled Analgesia Pump After Lumbar Spine Surgery
  Interventions: Drug: Oiceridine
- Sufentanil Group (Active Comparator): Sufentanil Patient-Controlled Analgesia Pump After Lumbar Spine Surgery
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — The postoperative PCA analgesia pump configuration plan is 1.5 μg/kg sufentanil diluted with saline to 100 ml.
  The specific parameters are a loading dose: 0.1 μg/kg sufentanil diluted with saline to 3 ml, administered 20-30 minutes before the end of surgery.
  Background infusion rate: 1.5 ml/h, PCA dose: 1 ml, lockout time: 10 minutes.
  Arms: Sufentanil Group
Drug: Oiceridine — The postoperative PCA analgesic pump regimen is 0.5 mg/kg of oliceridine diluted with saline to 100 ml. The specific parameters are a loading dose: 0.03 mg/kg of Oxycodone diluted with saline to 3 ml, administered 20-30 minutes before the end of surgery. Background infusion rate: 1.5 ml/h, PCA dose: 1 ml, lockout interval: 10 minutes.
  Arms: Oliceridine Group

SUMMARY:
Osemitidine fumarate is a novel G protein-biased ligand μ-opioid receptor agonist. Previous studies have confirmed its potent analgesic effects and safety: compared with morphine, it reduces respiratory depression and gastrointestinal dysfunction. This study aims to evaluate the effects of osemitidine on postoperative gastrointestinal function recovery and pain in patients undergoing lumbar spine surgery through a multicenter, double-blind, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old;
* Patients undergoing lumbar surgery under general anesthesia (within 3 segments) and expected to receive postoperative patient-controlled analgesia;
* ASA classification I-III;
* BMI between 18 and 30 kg/m²;
* Informed consent obtained from the patient.

Exclusion Criteria:

* Use of any painkillers within 3 days before surgery; or long-term treatment with non-steroidal anti-inflammatory drugs (NSAIDs), defined as: within 3 months before surgery, use of NSAIDs daily for more than 2 consecutive weeks;
* Presence of intestinal obstruction or suspicious symptoms: nausea and vomiting, abdominal bloating and pain, cessation of gas or bowel movements within the past two weeks, imaging suggesting intestinal dilation, or large amounts of air-fluid levels;
* Patients with severe liver dysfunction (based on Child-Pugh classification, grade C);
* History of or planned gastrointestinal surgery;
* Patients allergic to the study drug;
* Pregnant or breastfeeding patients;
* QTcF abnormalities, males >450 ms, females >470 ms;
* Participation in other drug trials within the past 30 days;
* Long-term use of opioids (defined as: within 12 months before surgery, use for more than 1 month, more than 3 days per week, with daily doses exceeding 15 mg morphine equivalent);
* Pre-existing neurological or psychiatric disorders: such as epilepsy, depression, schizophrenia, etc.;
* Patients deemed unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching the GI-3 composite endpoint within postoperative 24 hours | postoperative 24 hours
  Proportion of patients reaching the GI-3 composite endpoint (tolerating solid food and passing gas/bowel movement) within postoperative 24 hours

SECONDARY OUTCOMES:
Proportion of patients reaching the GI-3 composite endpoint within postoperative 48 hours | postoperative 48 hours
  Proportion of patients reaching the GI-3 composite endpoint (tolerating solid food and passing gas/bowel movement) within postoperative 48 hours
GI-3 | postoperative 48 hours
  GI-3: Reach the later of the following two milestones:
  ① Time of solid food tolerance: No vomiting occurs within 4 hours after eating food that requires chewing ;
  ② Time of first flatus or first bowel movement (whichever comes first).
IFEED score | postoperative 24 and 48 hours
  IFEED scores at postoperative 24 and 48 hours The I-FEED score is a novel outcome measure for POI, developed by expert consensus. It contains five elements (intake, response to nausea treatment, emesis, exam, and duration, each scored with 0, 1, or 3 points) and classifies patients into normal, postoperative gastrointestinal intolerance (POGI), and postoperative gastrointestinal dysfunction (POGD)(normal 0-2, POGI 3-5, POGD 6+ points)
Postoperative SPID | postoperative 24 and 48 hours
  Summed Pain Intensity Difference at postoperative 24 and 48 hours
Opioid consumption | postoperative 24 and 48 hours
  Opioid consumption at postoperative 24 and 48 hours
remedial analgesia | postoperative 48 hours
  Times of remedial analgesia at postoperative 48 hours

OTHER OUTCOMES:
Postoperative nausea and vomiting | posoperative 48 hours
  Incidence of nausea and vomiting within 48 hours after surgery, proportion of patients requiring rescue antiemetics within 48 hours, and the amount of rescue antiemetics used within 48 hours

IPD SHARING:
Plan to Share IPD: Undecided